CLINICAL TRIAL: NCT04825249
Title: A New Modified Suture Bridge Technique for Medium-sized Rotator Cuff Tears: Functional and Radiological Outcomes of a Prospective Study
Brief Title: A New Modified Suture Bridge Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zhangyi
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Rotator Cuff Tears
Keywords: rotator cuff tear， modified suture bridge technique
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Whereas patients and surgeons were aware of the group assignments, the outcome assessors and data analysts were remained blinded during the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The traditional suture bridge technique group (Experimental): For the TSB group, if the tear type is confirmed to be medium-sized during the operation, TSB technique will be performed
  Interventions: Procedure: traditional suture bridge technique
- The modified suture bridge technique group (Experimental): For the MSB group, if the tear type is confirmed to be medium-sized during the operation, TSB technique will be performed
  Interventions: Procedure: modified suture bridge technique

INTERVENTIONS:
Procedure: traditional suture bridge technique — (A) Limbs of the sutures from the medial anchor were passed through torn tendon (B) the suture limbs were tied in a horizontal mattress suture pattern (C) the lateral row pressed the free tails of the knotted line on the greater tubercle of the humerus (D) the effect after completion of the TSB technique
  Arms: The traditional suture bridge technique group
Procedure: modified suture bridge technique — (A) Limbs of the sutures from the medial anchor and 2 tendon sutures were passed through the same position of torn tendon (B) the lateral row pressed free tails of the two tendon lines on the greater tubercle of the humerus (C) after examination of sufficient tension and stable fixation, sutures of medial row was knotted (D) the effect after completion of the MSB technique
  Arms: The modified suture bridge technique group

SUMMARY:
We aimed to introduce a new modified suture bridge technique and report the clinical outcomes and radiological assessments of modified suture bridge technique for medium rotator cuff tears.

DETAILED DESCRIPTION:
Purpose: We aimed to introduce a new modified suture bridge technique and report the clinical outcomes and radiological assessments of modified suture bridge technique for medium rotator cuff tears.

Methods: We prospectively followed 50 consecutive patients with medium rotator cuff tears treated with the modified suture bridge (MSB) or traditional suture bridge technique (TSB) from December 2018 and December 2019. On the basis of preoperative findings and MRI performance, 26 patients underwent MSB repair whereas 24 underwent TSB repair. Range of shoulder motion, visual analog scale score (VAS score), University of California-Los Angeles score (UCLA score), Constant-Murley shoulder score (Constant score), American Shoulder and Elbow Surgeons score (ASES score) were assessed. Magnetic resonance imaging were performed preoperatively and at 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* (1) full-thickness medium tears (1-3cm) of primary supraspinatus (SSP) tendon was identified on preoperative MRI and intraoperative arthroscopy, (2) undesirable conservative treatment for 3 months, (3)completed follow-up of 12 months postoperatively and patients who adhered to the rehabilitation plan.

Exclusion Criteria:

* (1) previous shoulder surgery, (2) Other pathological changes that would need to be addressed at the time of arthroscopic surgery, such as rotator cuff tear involving the subscapular (SSC) tendon，biceps tendon injury, (3) failure to follow our postoperative rehabilitation protocol and patients without regular follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Cuff integrity grade of MRI assessment | at 12 months postoperatively
  Grade I: sufficient thickness of tendon; Grade II: sufficient thickness of tendon and partial high intensity within tendon; Grade III: insufficient thickness of tendon without discontinuity; Grade IV: slight discontinuity in 1 or 2 images of oblique coronal plane and sagittal plane; Grade V:obvious discontinuity of tendons in more than 2 images of both oblique coronal plane and sagittal plane.
Muscle atrophy grade of MRI assessment | at 12 months postoperatively
  Grade I: a ratio between 1.00 and 0.60 can be considered as normal or slightly atrophied; Grade II: values between 0.60 and 0.40 suggest moderate atrophy. Grade III: values below 0.40 indicate serious or severe atrophy.
Fatty degeneration grade of MRI assessment | at 12 months postoperatively
  Grade 0: completely normal muscle; Grade 1: muscle contains some fatty streaks; Grade 2: there is more muscle than fat; Grade 3: equal distribution of fat and muscle; grade 4: more fat was present than muscle. Among them, grade 0 is normal, grade 1 and 2 are considered moderate, grade 3 and 4 are classified as severe.
Range of shoulder motion | at 12 months postoperatively
  Different range of motion of shoulder joint
The Visual Analog Scale score | preoperatively
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | at 12 months postoperatively
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
University of California-Los Angeles score | preoperatively
  The score mainly consists of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint mobility and muscle strength. Possible scores range from 0 to 35, a higher score means a better result.
University of California-Los Angeles score | at 12 months postoperatively
  The score mainly consists of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint mobility and muscle strength. Possible scores range from 0 to 35, a higher score means a better result.

SECONDARY OUTCOMES:
Constant-Murray Shoulder score | preoperatively
  An assessment method often used by orthopedic surgeons when assessing the condition of patients with shoulder joints.Possible scores range from 0 to 100#a higher score means a better result.
Constant-Murray Shoulder score | at 12 months postoperatively
  An assessment method often used by orthopedic surgeons when assessing the condition of patients with shoulder joints.Possible scores range from 0 to 100#a higher score means a better result.
American Shoulder and Elbow Surgeon score | preoperatively
  The evaluation criteria used to assess shoulder joint function based on the patients' pain and accumulated daily activities. Possible scores range from 0 to 100. The higher the score, the better the shoulder joint function.
American Shoulder and Elbow Surgeon score | at 12 months postoperatively
  The evaluation criteria used to assess shoulder joint function based on the patients' pain and accumulated daily activities. Possible scores range from 0 to 100. The higher the score, the better the shoulder joint function.

CONTACTS AND LOCATIONS:
Overall Officials: Tengbo Yu, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Shangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Proposals should be directed to zhangsports2021@sina.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website
URL: http://www.medresman.org.cn/uc/sindex.aspx

REFERENCES:
- [Result] Takeuchi Y, Sugaya H, Takahashi N, Matsuki K, Tokai M, Morioka T, Ueda Y, Hoshika S. Repair Integrity and Retear Pattern After Arthroscopic Medial Knot-Tying After Suture-Bridge Lateral Row Rotator Cuff Repair. Am J Sports Med. 2020 Aug;48(10):2510-2517. doi: 10.1177/0363546520934786. Epub 2020 Jul 14. PMID 32663065
- [Result] Kim KC, Shin HD, Lee WY, Yeon KW, Han SC. Clinical outcomes and repair integrity of arthroscopic rotator cuff repair using suture-bridge technique with or without medial tying: prospective comparative study. J Orthop Surg Res. 2018 Aug 28;13(1):212. doi: 10.1186/s13018-018-0921-z. PMID 30153852
- [Result] Dukan R, Ledinot P, Donadio J, Boyer P. Arthroscopic Rotator Cuff Repair With a Knotless Suture Bridge Technique: Functional and Radiological Outcomes After a Minimum Follow-Up of 5 Years. Arthroscopy. 2019 Jul;35(7):2003-2011. doi: 10.1016/j.arthro.2019.02.028. Epub 2019 May 27. PMID 31147110